CLINICAL TRIAL: NCT06279403
Title: Upfront Toripalimab Plus Axitinib Combined With Deferred Cytoreductive Nephrectomy for Metastatic Renal Cell Carcinoma
Brief Title: Upfront Immune Checkpoint Inhibitors With Deferred Cytoreductive Nephrectomy for Metastatic Renal Cell Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2023-0277
Record Dates: First submitted 2024-01-29; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Clear-cell Metastatic Renal Cell Carcinoma; Immune Checkpoint Inhibitors; Cytoreductive Nephrectomy
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma | interventions — toripalimab; Axitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Experimental arm
  Interventions: Drug: Toripalimab; Procedure: Cytoreductive Nephrectomy; Drug: Axitinib

INTERVENTIONS:
Drug: Toripalimab — Preoperative Treatment with Toripalimab: Administer 240mg of Toripalimab via intravenous infusion every 3 weeks for a total of 4 cycles.
Procedure: Cytoreductive Nephrectomy — Radical Nephrectomy: Complete resection of the tumor and affected kidney within the renal fascia.
  Partial Nephrectomy: Complete resection of the tumor while preserving maximal kidney function.
  Lymph Node Dissection: For patients with evident enlargement of retroperitoneal lymph nodes preoperatively, perform lymph node dissection at the renal hilum, along the ipsilateral major vessels, and anterior to the ipsilateral major vessels. Lymph node dissection is not required for patients without evident enlargement of retroperitoneal lymph nodes preoperatively.
Drug: Axitinib — Preoperative Treatment with Axitinib: Administer 5mg of axitinib orally twice daily for a duration of 3 months.

SUMMARY:
Study Objective: To determine the efficacy of upfront immune checkpoint inhibitors combined with deferred cytoreductive nephrectomy in treating metastatic renal cell carcinoma.

Primary Endpoint: Pathological Major Response (MPR), defined as the percentage of residual tumor cells <10% in the primary tumor after nephrectomy.

Study Design:

Population: Participants meeting the diagnostic criteria with biopsy-proven clear cell renal cell carcinoma, IMDC score ≤3, or ≤5 metastatic lesions involving ≤3 organs.

Sample Size: 20 participants.

Patient Grouping: Non-randomized.

Interventions: Eligible participants will receive upfront treatment with a combination of Axitinib and Toripalimab for 4 cycles. After 2 cycles of treatment, radiological assessment will be conducted using RECIST 1.1 criteria. If disease progression is observed, the clinical trial will be terminated, and second-line treatment will be initiated according to guidelines. If disease progression is not observed, treatment will continue for 2 additional cycles followed by repeat radiological assessment before undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

Voluntary consent to participate in this study and signing of an informed consent form.

Male or female participants aged ≥18 years and <80 years. Histologically diagnosed with clear cell carcinoma or predominantly clear cell renal cell carcinoma.

Clinical stage determined by CT or MRI: anyTN1M0 or anyTN0M1; IMDC score ≤3, or ≤5 metastatic lesions involving ≤3 organs; and the primary tumor (unilateral or bilateral) is resectable.

ECOG performance status: 0 or 1. No clinically significant cardiac, bone marrow, hepatic, or renal function abnormalities.

A willingness and ability to comply with testing and follow-up procedures.

Exclusion Criteria:

Non-clear cell carcinoma. Severe liver or kidney dysfunction, or other severe diseases. Immune deficiency, organ transplantation, or autoimmune diseases. Severe central nervous system diseases. Other malignant tumors within the past 5 years, except for cured basal cell carcinoma of the skin and cervical carcinoma in situ.

Unable to comply with regular follow-up visits due to psychological, social, family, or geographical reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Major Response (MPR) | through study completion, an average of 1 year
  The percentage of residual tumor cells in the primary tumor after surgery, with MPR defined as less than 10% of residual tumor cells in the pathology report.

IPD SHARING:
Plan to Share IPD: No